CLINICAL TRIAL: NCT01386801
Title: Multicenter Research Study to Build a Repository That Will Allow Researchers to Study Chronic Diseases in the Population of Central Indiana
Brief Title: Multicenter Research Study to Build a Repository to Study Chronic Diseases in Indiana
Acronym: IHS
Status: Active, not recruiting | Type: Observational
Sponsor: Fairbanks Institute (Other)
Collaborators: Indiana University School of Medicine (Other); Richard M. Fairbanks Foundation (Other); BioCrossroads (Other); Regenstrief Institute, Inc. (Other)
Responsible Party: Cynthia Helphingstine, Fairbanks Institute for Healthy Communities
Other Study IDs: FIHC-2009-01
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus Type II
Keywords: Diabetes; Controls; Biospecimen
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA = 1 Serum = 2 Plasma = 2 RNA = 2
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- People with Diabetes Mellitus Type II: 500 subjects will have T2D
- Healthy: 500 persons who do not have T2D, hypertension or hypercholesterol

SUMMARY:
Blood samples and health information (e.g., age at diagnosis, test results) are collected for the purposes of genetic research. The blood samples are assigned a number and stored in a repository for safe keeping until they are needed for a research project. Participants are persons who are healthy (not having high blood pressure, diabetes, or high cholesterol levels) or persons who have Diabetes Mellitus Type II(T2D) and live in Indiana. Participants complete a questionnaire at the time the blood sample is drawn. Visits are repeated at 2 and 5 years after initial contact. Researchers apply to the Fairbanks Institute for use of the blood samples and health information minus participant names and contact information. Their research is required to be related to find genes or substances made by genes that may be involved in Diabetes Mellitus Type II with the purpose of improving the investigators understanding of the illness potentially leading to the development of new diagnostic tools for identifying the illness, new treatments,or preventative measures.

DETAILED DESCRIPTION:
Study Aim:

The purpose of this study is to create an extensively annotated bio-repository platform for hypothesis-driven research that will lead to advancements in the diagnosis, treatment and prevention of diseases common to the population of Indiana. The second phase of this research platform will be created by collecting blood samples from two groups of individuals in the Central Indiana community, one with documented evidence of Diabetes Mellitus Type II(T2D), and a second group of age, gender and ethnicity matched individuals without clinical evidence of Diabetes. Each individual's blood sample will be linked to their clinical, demographic and epidemiological information, gathered both retrospectively and prospectively.

Recruitment:

This study will include 500 individuals with T2D (the T2D Group) and 500 individuals who are age, gender, and ethnicity matched to the T2D Group, but without presentation of clinical evidence of T2D (the Control Group). To reflect the growing representation of Hispanics in Central Indiana, Hispanics will be overly recruited in both groups so that the study population accurately reflects the general population of Central Indiana.

Follow-up:

As this is a prospective, longitudinal study, follow-up of study subjects is intended to include two follow up visit and continue indefinitely, unless, of course, at any time, consent for further follow-up is withdrawn by the subject. Follow-up will include visits at 2 and 5 years post initial contact and continuing access to the subject's medical record to pursue data concerning changes in the subject's health. Subjects may be contacted by telephone, mail or email every twelve months to ask if they wish to continue participation in the study. The 2 and 5 year follow up visits mirror the initial visit.

The collected dataset (made up of the collected blood samples linked to clinical and epidemiological information collected retrospectively and prospectively), will be used in medical research to find genes, or gene products such as RNA or proteins that will help in understanding the causes of disease and will guide the development of new treatments

ELIGIBILITY:
Inclusion Criteria:T2D Group

Study subjects will be recruited for the T2D group based on a history confirmed by the medical record of at least one of the following:

* A fasting blood glucose of greater than or equal to 126 mg/dL on two separate occasions
* A random (non-fasting) blood glucose of greater than or equal to 200 mg/dL on two separate occasions
* A blood glucose of greater than 200 mg/dL at 2 hours during a standard oral glucose tolerance test
* A HgbA1c of greater than or equal to 6.5%

Females who are pregnant will be excluded.

Control Group

Study subjects for the Control Group will have:

* no confirmed history of T2D as defined above
* A fasting blood glucose of 100 mg/dL or less

Medical records will be obtained to ensure subjects meet study inclusion criteria.

-

Exclusion Criteria:Exclusion criteria for both the T2D Group and the Control Group are a known or reported history of:

* Hepatitis B
* Hepatitis C
* AIDS (HIV positive)
* Tuberculosis
* Cancer (including melanoma, but excluding low-malignancy skin cancer)
* Non-autologous bone marrow transplant
* Blood transfusion within 120 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living in the state of Indiana
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-12; Primary Completion 2049-12 (Estimated); Study Completion 2050-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anantha Shekhar, MD, Principal Investigator — Indiana University School of Medine/CTSI
Locations (11):
- United States (11):
  - American Health Network, Avon, Indiana
  - Investigator's Research Group, Brownsburg, Indiana
  - American Health Network, Franklin, Indiana
  - American Health Network, Greenfield, Indiana
  - American Health Network, Indianapolis, Indiana
  - Krannert Cardiology, Indianapolis, Indiana
  - Oral Health Research Institute, Indianapolis, Indiana
  - IU School of Medicine/CTSI, Indianapolis (Downtown), Indiana
  - Alivio Medical Center, Indianapolis (Spanish Speaking), Indiana
  - IU Medical Group, Indianapolis (Spanish/English Speaking), Indiana
  - American Health Network, Muncie, Indiana

REFERENCES:
- See also: Accelerated Clinical and Translational Research — http://www.indianactsi.org/